CLINICAL TRIAL: NCT04637100
Title: Effect of Free Mobile or Tablet-based Applications on Stroke-Related Cognitive Impairment in Inpatient Rehabilitation
Brief Title: Gaming Apps Post-Stroke
Acronym: GAPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in research personnel
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Christopher Tarver, Assistant Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5200471
Record Dates: First submitted 2020-11-03; First posted 2020-11-19 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Stroke; Cognitive Impairment; Executive Dysfunction; Cognitive Change; Cognitive Deficit
Keywords: Stroke; cerebrovascular accident
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The patient will utilize their personal mobile or tablet device to play a pre-selected set of problem-solving games for a goal of 1 hour daily for the duration of their inpatient rehabilitation stay (approximately 3 weeks).
  Interventions: Other: Mobile or tablet-based gaming applications
- Control (Active Comparator): The patient will utilize their personal mobile or tablet device to watch a pre-selected set of stroke-related educational videos for a goal of 1 hour daily for the duration of their inpatient rehabilitation stay (approximately 3 weeks).
  Interventions: Other: Stroke-related educational videos

INTERVENTIONS:
Other: Mobile or tablet-based gaming applications — Subject will use their own personal smartphone or tablet device to play from a collection of pre-selected gaming applications. The collection is made of puzzle-type games available on both Android and iOS without excessive ads and with clear or self-explanatory instructions. Subject will be instructed to play for 1 hour daily for the duration of their acute inpatient rehabilitation stay (approximately 3 weeks).
  Arms: Experimental
Other: Stroke-related educational videos — Subject will use their own personal smartphone or tablet device to watch videos from a collection of pre-selected educational videos. These include topics on stroke recognition, stroke recovery process, patient experiences with stroke, rehabilitation after stroke, activities of daily living equipment instructions. Subject will be instructed to watch for 1 hour daily for the duration of their acute inpatient rehabilitation stay (approximately 3 weeks).
  Arms: Control

SUMMARY:
The investigators aim to explore the effect of puzzle mobile or tablet-based games on problem-solving impairment resulting from a first-time stroke. This is a randomized-controlled trial with the intervention arm consisting of puzzle gaming applications and the control arm consisting of stroke-relevant educational videos provided and encouraged throughout the course of participants' acute inpatient rehabilitation stay.

DETAILED DESCRIPTION:
Study subjects will be randomized to a control or experimental group and allocation will be concealed. The experimental group will consist of the subject utilizing their personal mobile or tablet device to play a pre-selected set of problem-solving games for a goal of 1 hour daily. The control group will utilize their personal mobile or tablet device to perform the non-problem-solving task of watching educational videos of their choice from a pre-selected set of videos for the same amount of time daily. The intervention gaming arm will be provided different gaming apps if they lose interest or find a particular game too easy or too difficult. The control video arm will be provided different educational videos according to their needs that may change throughout their inpatient stay.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-89
2. Hospitalized at Loma Linda East Campus Rehabilitation Hospital
3. First time stroke patient
4. mild to moderate problem-solving impairment without severe deficit in any other cognitive domain on admission speech evaluation
5. Have daily access while inpatient to a personally owned Apple or Android smartphone or tablet device prior to the initial session.

Exclusion Criteria:

1. Unable to understand and follow verbal and written instructions in English
2. Presence of aphasia that limits device use or ability to provide consent
3. Presence of pre-stroke speech, language, or cognitive disorder
4. Unable to operate device due to cognitive, physical, or visual impairment

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Scales of Cognitive and Communicative Ability for Neurorehabilitation (SCCAN) | From date of randomization until the day of discharge, assessed at beginning and end of this period, up to 5 weeks
  Assesses cognitive-communicative deficits and functional ability in patients in rehabilitation hospitals, clinics, and skilled nursing facilities. The SCCAN contents relate to daily activities that adults would be expected to perform for independent living. The SCCAN has eight scales and a total score:
  Oral Expression, Orientation, Memory, Speech Comprehension, Reading Comprehension, Writing, Attention, Problem Solving
  Typical functioning = 87-94 Mild impairment = 69-86 Moderate impairment = 47-68 Severe impairment = 0-46

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | From date of randomization until the day of discharge, assessed at beginning and end of this period, up to 5 weeks
  Rapid screen of cognitive abilities designed to detect mild cognitive dysfunction consisting of 16 items and 11 categories assessing multiple cognitive domains
  No cognitive impairment >=25 Mild cognitive impairment = 20-24 Severe cognitive impairment < 20
Modified Gaming Engagement Questionnaire | From date of randomization until the day of discharge, assessed at end of this period, up to 5 weeks. Qualitative feedback only.
  15-item questionnaire for feedback on engagement during game-playing or video watching
Program Evaluation | From date of randomization until the day of discharge, assessed at end of this period, up to 5 weeks. Qualitative feedback only.
  11 item questionnaire for feedback on participant experience

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Tarver, MD, Principal Investigator — Loma Linda University
Locations (1):
- Tom and Vi Zapara Rehabilitation Pavilion, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No